CLINICAL TRIAL: NCT00434317
Title: A Multicenter, Open-label Study to Determine the Effect of iv. Zoledronic Acid on Pain and Quality of Life in Patients With Bone Metastases With or Without Skeletal Related Events (SRE) Resulting From Breast Cancer and Prostate Cancer
Brief Title: Assessment of Pain and Quality of Life in Breast and Prostate Cancer Patients With Bone Metastases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EHU03
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Neoplasm Metastasis
Keywords: Metastasis; Neoplasm; pain; breast cancer; prostate cancer; bone metastasis
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Pain; Breast Neoplasms; Prostatic Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- ZOL446 (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of zoledronic acid administered intravenously every 3-4 weeks in patients with bone metastases from either breast cancer or prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* Ambulatory patients >18 years
* Proof of breast cancer or prostate cancer
* Diagnosis of at least one cancer-related bone lesion that is detectable on conventional radiographs or bone scan at screening
* Negative pregnancy test
* ECOG performance status of 0,1 or 2

Exclusion criteria:

* Patients with abnormal renal function
* Patients with clinically symptomatic brain metastases
* Known hypersensitivity on zoledronic acid or other bisphosphonates
* Pregnancy or lactation

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-08; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Measurement of pain assessed by a Visual Analogue Scale (VAS) | throughout the study

SECONDARY OUTCOMES:
Quality of Life assessment at baseline and last visit | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Székesfehérvár